CLINICAL TRIAL: NCT01927614
Title: Advanced Cardiac Imaging in Cardiac Allograft Vasculopathy
Status: Terminated | Type: Observational
Why Stopped: PI resigned from the department of medicine, dalhousie university and the nova scotia health authority effective august 24 2015
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: CDHA_CAV
Record Dates: First submitted 2013-08-12; First posted 2013-08-22 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-10

CONDITIONS: Heart Transplantation
Keywords: Cardiac Allograft Vasculopathy; Cardiac MRI; Cardiac CT; Observational study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: 20 patients 1-year post heart transplant will undergo standard of care invasive cardiac catheterization but will also have intravascular ultrasound performed to measure the maximal intimal thickness of the proximal left anterior descending artery. Patients will be dichotomized into those with MIT <0.5mm (10 patients) and those with MIT >0.5mm (10 patients). All 20 patients will undergo both cardiac CT and cardiac MRI with perfusion imaging.
  Interventions: Radiation: Cardiac CT
- Cohort 2: 10 patients 1 year post heart transplant classified as CAV grade 0 by standard cardiac catheterization will undergo both cardiac CT and cardiac MRI with perfusion imaging.
  Interventions: Radiation: Cardiac CT
- Cohort 3: 10 patients with a diagnosis of CAV grade 1 as assessed by routine coronary angiogram at any time point post heart transplantation, will undergo cardiac CT and cardiac MRI with perfusion imaging
  Interventions: Radiation: Cardiac CT

INTERVENTIONS:
Radiation: Cardiac CT — A 128-slice dual-source CT system will be used (Somatom Definition Flash, Siemens Healthcare, Germany).
  The CT scan protocol will comprise 3 steps.
  1. Prospectively gated calcium scoring.
  2. Stress-myocardial CT perfusion.
  3. Rest Coronary CT angiography and myocardial CT perfusion. Automated computed tomography dose index (CTDIvol) and dose- length-product (DLP) will be collected from the scanner, and effective dose will be calculated using the DLP conversion factor (0.014) for each component of the cardiac CT protocol. Based on local dose audits the predicted dose range will be 3.5 mSv to 8 mSv depending on patient body habitus.

SUMMARY:
Cardiac allograft vasculopathy (CAV) is a process of both immune and non-immune mediated thickening of the heart arteries of transplanted hearts. CAV limits the long term survival of heart transplant patients and is one of the common causes of death in the late post transplant period. Current methods of detecting CAV rest with invasive cardiac catheterization which carry repeated risks, as this test needs to be performed periodically through the life of a heart transplant patient. Traditional methods of coronary angiography identify CAV late in its course and is a crude method of evaluating coronary anatomy in heart transplant patients. Intravascular ultrasound is an additive tool that is able to detect early CAV before it becomes angiographically apparent, but still requires invasive cardiac catheterization to perform. However, it also limits assessment to the major epicardial arteries and does not give any information regarding the smaller branch vessels and cardiac microvasculature. Advances in cardiac CT and cardiac MRI hold potential to evaluate for CAV non-invasively. In addition, perfusion techniques may provide additional functional information regarding the status of the microvascular.

In this pilot study, we aim to demonstrate the feasibility of cardiac CT and cardiac MRI with and without perfusion protocols, in patients post-heart transplant and to describe and compare CT and MRI findings in patients with established CAV versus those with no CAV, as diagnosed by standard invasive methods.

DETAILED DESCRIPTION:
Heart transplantation is a viable treatment option for select patients with end-stage heart failure, with 1-year survival rates for heart transplantation approximating 85%. Of those who survive the first year, >90% are alive at 5 years. In the early post-transplant period, rejection of the donor heart due to activation of the recipients immune system, is the most worrisome complication and most common cause of morbidity and mortality. With time, the risk of rejection declines and cardiac allograft vasculopathy (CAV) represents the most common cause of heart failure and death in heart transplant recipients. CAV is a form of coronary artery disease in the transplanted heart. It develops due to a variety of immune and non-immune mediated mechanisms. It differs significantly from coronary artery disease in normal hearts, in that it affects arteries of all sizes (not just the main arteries visible by coronary angiography) and it involves thickening of the inner layer of the arteries, rather than the surface lining of the arteries as in traditional coronary artery disease. Early CAV is clinically silent. Patients are most often diagnosed by routine coronary angiographic surveillance (standard of care), or by declining heart function by surveillance imaging (standard of care), with no evidence of any organ rejection.

Coronary angiography and assessment of heart function remain the cornerstone for diagnosis of CAV. The main limitation of angiography is its inability to identify mild or early disease, as an apparently normal angiogram can underestimate the presence of CAV. Intra-vascular ultrasound (IVUS) at coronary angiography has been evaluted as an adjunctive mordality for assessing and diagnosing early CAV. Certain IVUS parameters have been correlated with high risk for development of CAV and overall worse prognosis long term.

Detection of CAV has important therapeutic and prognostic implications. Once detected by angiography, the likelihood of progression to severe CAV within 5 years is 19%. The overall likelihood of death or re-transplantation as a result of CAV is approximately 50% for severe CAV. Changes are made to medical therapy targeted at slowing or halting CAV progression and patients are evaluated for re-transplantation sooner rather than later, depending on the rate of progression.

Currently, CAV is diagnosed by cardiac catheterization performed at routine intervals post transplant, with or without the use of IVUS. This is an invasive test with complications including bleeding, vascular damage, renal failure, stroke, heart attack or death. It has low sensitivity for identifying early CAV. Recent advances in cardiac magnetic resonance imaging (CMR) and cardiac CT imaging (CCT) present a unique opportunity to investigate these non-invasive modalities in CAV. To date, there are no studies in this field.

We propose to evaluate whether functional CCT and/or CMR perfusion abnormalities, calcium scoring by CCT, and late gadolinium enhancement by CMR, is feasible in heart transplant patients and whether these modalities can detect abnormalities that correlate to cardiac catheterization results and detect early CAV before it becomes angiographically apparent. This pilot study will be the first of its kind in the heart transplant population. We aim to demonstrate feasibility and safety of CCT/CMR in heart transplant patients and correlate specific CMR/CCT abnormalities to established angiographic apparent CAV. This will allow further prospective evaluation of this exciting non-invasive modality in CAV detection with larger research studies by our group.

The clinical implications are significant in that we may reduce the number of invasive procedures performed and identify CAV earlier, leading to the institution of earlier therapies, such as proliferation signal inhibitors, that may alter the natural history of this disease in effort to prolong the life of the transplanted heart.

Specific Objectives:

Primary Objectives:

1. The number of patients with adverse events from CCT and CMR
2. Determine recruitment rates for future studies, logistics of testing, and the ability to perform the tests

Secondary Objectives:

1. Describe the CCT and CMR imaging findings in CAV

   1. Identify and describe structural and functional CMR abnormalities in established angiographically apparent CAV using novel imaging protocols, including stress-rest perfusion imaging.
   2. Identify and describe structural and functional cardiac CT abnormalities in established angiographically apparent CAV using novel imaging protocols, including stress-rest perfusion imaging.
2. Correlation between intimal thickening by IVUS imaging at cardiac catheterization and CCT/CMR perfusion abnormalities at one year post heart transplant.
3. Correlation between CCT/CMR perfusion abnormalities at one year post heart transplant with the development of angiographically apparent CAV, graft dysfunction, cardiac adverse events, and overall survival long term, and compare CCT to CMR in this regard (Cohort 1 & 2 below)

Study Design: Patients will be recruited into 1 of 3 cohorts from the heart transplant program at the QE II Health Science Center, Halifax Infirmary site, using a protocol approved by the institutional research ethics board. Eligible patients are those scheduled for routine invasive coronary angiography, > 18 years of age, > 12 months post-transplant and be able to undergo both CCT and CMR. Exclusion criteria include a creatinine clearance (CrCl) calculated < 45ml/min, contraindications or inability to administer intravenous beta-blockers or calcium channel blockers and standard contraindications to CMR, contrast media, and adenosine. Patients will be identified by Dr. Brian Clarke who is involved the care of all heart transplant patients at the QE II Health Science Centre

Data will be analyzed as follows:

1. Feasibility will be determined based on successful rate of recruitment and completion of CCT/CMR scans in cohort 3.
2. Patients eligible for cohort 3 require the diagnosis of CAV 1 at any time point post-transplant. The attending transplant cardiologist involved makes this assessment. More advanced CAV is excluded. These patients will be analyzed without a comparator group. For CCT, calcium scoring, intimal thickening, and perfusion abnormalities will be described and analyzed for their correlation to angiographic findings. CMR imaging will describe late gadolinium enhancement, structural changes, and perfusion abnormalities and be analyzed for their correlation to angiographic findings. In a separate analysis, these patients will also be compared with those in cohort 2 to determine the non-invasive imaging differences between CAV1 and CAV0 patients.
3. Cohort 1 will be analyzed separately; comparing those with MIT <0.5mm to those with MIT > 0.5mm for differences in CCT/CMR imaging and perfusion abnormalities. CCT will be compared with CMR in both MIT subgroups. We anticipate to identify perfusion abnormalities in the MIT > 0.5mm group and no perfusion abnormalities in the MIT < 0.5mm. Patients in cohort 1 will be followed long term for the development of angiographically apparent CAV, adverse cardiac events, graft dysfunction, and death.

Results will be reported mainly in a descriptive manner, so that data will be summarized in percentage, mean or median, where applicable.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Greater than or equal to 12 months post transplant
* Able to undergo cardiac CT and cardiac MRI

Exclusion Criteria:

* Creatinine clearance less than or equal to 45ml/min per 1.73m2)
* Severe aortic stenosis
* Long-QT syndrome (corrected QT >440ms)
* AV block grade II/III
* Sick sinus syndrome
* New York Heart Association heart failure class III/IV
* Chronic obstructive pulmonary disease
* Asthma
* Atrial fibrillation
* Left ventricular ejection fraction <50%
* Presence of a pacemaker or ICD
* Presence of any metal in body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Transplant Patients
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-10-13 (Actual); Primary Completion 2015-07-17 (Actual); Study Completion 2015-07-17 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events from cardiac CT and cardiac MRI scan in heart transplant patients | Day 1
  Testing the safety and feasibility of performing cardiac CT and MRI with perfusion protocols in heart transplant patients. Adverse events: serum creatinine increase >25% from baseline within 1 week, drop in systolic blood pressure >30mmHg, arrhythmias, chest pain, shortness of breath during drug infusion for perfusion protocols, inability to reduce heart rate <80bpm for cardiac CT.

SECONDARY OUTCOMES:
Describe CT and MRI imaging findings of established CAV | Day 1
Correlation between intimal thickening by IVUS imaging at cardiac catheterization and CCT and CMR perfusion abnormalities | Day 1
The association between CCT/CMR perfusion abnormalities one year post transplant and the development of angiographically apparent CAV, graft dysfunction, cardiac adverse events, and overall survival long term | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Clarke, MD, Principal Investigator — Staff Cardiologist and Clinical Assistant Professor, Division of Cardiology, QE II Health Science Centre, Dalhousie University and Capital District Health Authority
Locations (1):
- Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia, Canada